CLINICAL TRIAL: NCT00004011
Title: A Randomized Phase III Trial of Surgery Alone or Surgery Plus Preoperative Paclitaxel/Carboplatin in Clinical Stage IB (T2N0), II (T1-2N1, T3N0) and Selected IIIA (T3N1) Non-Small Cell Lung Cancer (NSCLC)
Brief Title: S9900: Surgery With or Without Combination Chemotherapy in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067223; S9900 (Other: SWOG); S9900 (Other: ECOG); S9900 (Other: NCCTG); RTOG-L0015 (Other: RTOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preooperative chemo followed by surgery (Experimental): carboplatin paclitaxel conventional surgery
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery
- Surgery alone (Active Comparator): conventional surgery
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Drug: carboplatin
  Arms: preooperative chemo followed by surgery
Drug: paclitaxel
  Arms: preooperative chemo followed by surgery
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if surgery plus combination chemotherapy is more effective than surgery alone for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival of patients with previously untreated stage IB, II, or selected IIIA non-small cell lung cancer after preoperative chemotherapy comprising paclitaxel and carboplatin plus surgery vs surgery alone.
* Compare these regimens in terms of operative mortality and other toxic effects in these patients.
* Evaluate the response rates (confirmed and unconfirmed) and toxic effects associated with combined paclitaxel and carboplatin in these patients.
* Obtain samples for correlation of radiologic, pathologic, molecular, and biologic factors with the outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to clinical stage (IB or IIA vs IIB or IIIA).

Patients are randomized to one of two treatment arms:

* Arm I: Patients undergo thoracotomy. All accessible hilar (level 10) lymph nodes are dissected, and complete mediastinal lymph node sampling is performed.
* Arm II: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for a maximum of 3 courses in the absence of disease progression or unacceptable toxicity. Within 2-6 weeks of course 3, patients undergo thoracotomy and lymph node dissection as in arm I.

Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually until year 10.

PROJECTED ACCRUAL: A total of 600 patients (300 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven non-small cell lung cancer (NSCLC), meeting 1 of the following staging criteria:

  * Stage IB (T2, N0)
  * Stage II

    * T1-2, N1 with negative mediastinoscopy OR
    * T3, N0
  * Selected stage IIIA with negative mediastinoscopies

    * T3, N1, excluding superior sulcus
    * Positive level 10 hilar nodes allowed if mediastinoscopy negative
* Apical tumors with no clinical symptoms allowed
* No symptomatic tumors (T3, N0 or T3, N1) involving the superior sulcus

  * No Pancoast's tumors
* Negative mediastinoscopy required in all patients with clinically positive mediastinal or hilar lymph nodes to ensure no N2 disease
* Bidimensionally measurable or evaluable disease by chest x-ray or contrast-enhanced CT scan

  * T3, N0 disease assessable only by bronchoscopy must be affirmed by 2 observers and documented by photograph that includes main carina

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* WBC at least 4,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min

Pulmonary:

* See Disease Characteristics
* Preresection FEV_1 greater than 2.0 L OR
* Predicted postresection FEV_1 greater than 1.0 L
* No postobstructive pneumonia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious infection
* No other serious medical condition that would preclude study compliance
* No prior allergic reactions to drugs containing Cremophor
* No prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior systemic radiotherapy for NSCLC
* No concurrent radiotherapy

Surgery:

* At least 5 years since prior resection of lung disease

Other:

* No other concurrent investigational therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 1999-10; Primary Completion 2005-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Bunn, MD, Study Chair — University of Colorado, Denver; Joseph A. Treat, MD, Study Chair — Fox Chase Cancer Center; Randolph S. Marks, MD, Study Chair — Mayo Clinic; Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (287):
- United States (267):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Montgomery Cancer Center, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Centers - Sacramento, Sacramento, California
  - Radiation Medical Group, Incorporated, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of St. Raphael, New Haven, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Halifax Medical Center, Daytona Beach, Florida
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Scott and White Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Radiation Oncology Center at Caritas Regional Cancer Center, Louisville, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - NSMC Cancer Center, Peabody, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Medical Center of Princeton, Princeton, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Cancer Center at Christ Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Frank C. Love Cancer Institute at St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes-Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre at Regional Hospital of Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Pisters KM, Vallieres E, Crowley JJ, Franklin WA, Bunn PA Jr, Ginsberg RJ, Putnam JB Jr, Chansky K, Gandara D. Surgery with or without preoperative paclitaxel and carboplatin in early-stage non-small-cell lung cancer: Southwest Oncology Group Trial S9900, an intergroup, randomized, phase III trial. J Clin Oncol. 2010 Apr 10;28(11):1843-9. doi: 10.1200/JCO.2009.26.1685. Epub 2010 Mar 15. PMID 20231678
- [Result] Pisters K, Vallieres E, Bunn PA, et al.: S9900: surgery alone or surgery plus induction (ind) paclitaxel/carboplatin (PC) chemotherapy in early stage non-small cell lung cancer (NSCLC): follow-up on a phase III trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-7520, 389s, 2007.
- [Result] Pisters K, Vallieres E, Bunn P, et al.: S9900: a phase III trial of surgery alone or surgery plus preoperative (preop) paclitaxel/carboplatin (PC) chemotherapy in early stage non-small cell lung cancer (NSCLC): preliminary results. [Abstract] J Clin Oncol 23 (Suppl 16): A-LBA7012, 624s, 2005.